CLINICAL TRIAL: NCT02138578
Title: A Phase II Randomized Trial Comparing Stereotactic Body Radiation Therapy to Radiofrequency Ablation for the Treatment of Localized Renal Cell Carcinoma (RCC)
Brief Title: Trial Comparing Stereotactic Body Radiation Therapy to Radiofrequency Ablation for Renal Cell Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to changes in scanning procedure, and infeasible biopsy and baseline imaging, the trial closed for poor accrual and inability to follow patients.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2013.069; HUM00076618 (Other: University of Michigan)
Record Dates: First submitted 2014-04-16; First posted 2014-05-14 (Estimated); Results first posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-10

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Radiosurgery; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Randomized SBRT (Experimental): Patients who meet eligibility criteria (unilateral primary renal cell carcinoma less than 4 cm in greatest diameter) and are randomized to Stereotactic Body Radiation Therapy (SBRT) will receive SBRT delivered in fractions of 20 Gy, approximately every other day, for a total of three treatments. If the target is deemed too close to organs at risk, 5 fractions of up to 10 Gy per fraction will be prescribed.
  Interventions: Radiation: SBRT
- Randomized RFA (Active Comparator): Patients who meet eligibility criteria (unilateral primary renal cell carcinoma less than 4 cm in greatest diameter) and are randomized to Radiofrequency Ablation (RFA) will receive RFA.
  Interventions: Radiation: RFA
- Non-Randomized SBRT (Active Comparator): Patients with renal cell carcinoma's greater than or equal to 4 cm in diameter, and up to 8 cm in diameter, may be placed in the non-randomized stereotactic body radiation therapy arm. Patients with tumors not amenable to RFA, those with metastatic disease, and those who elect a noninvasive means of treatment will also be eligible to receive treatment in the non-randomized SBRT cohort.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT
  Other Names: Stereotactic Body Radiation Therapy
  Arms: Non-Randomized SBRT; Randomized SBRT
Radiation: RFA
  Other Names: Radiofrequency Ablation
  Arms: Randomized RFA

SUMMARY:
This study will assess whether Stereotactic Body Radiation Therapy (SBRT) can provide comparable local control, with similar or improved toxicity rates compared to Radio Frequency Ablation (RFA) when treating small renal cell carcinomas.

ELIGIBILITY:
Inclusion Criteria for SBRT vs. RFA Randomization:

* Patients with renal cell carcinoma less than 4 cm in maximum diameter, who are poor surgical candidates are eligible for randomization between SBRT and RFA (Renal cell carcinoma must be pathologically proven).
* The primary tumor must be in a location amendable to RFA within the kidney.
* Patients must be appropriate candidates for RFA, with platelets ≥50,000/mm3 and an international normalized ratio of 1.5.
* Patients must have an ECOG (a measurement of general well being and activities of daily living; scores range from 0 to 5 where 0 represents perfect health) score ≤ 3.
* There is no required minimum renal function (patients will be counseled about the possible need for dialysis, if applicable, just as would be the case for radical or partial nephrectomy).
* Patients must sign an informed consent form approved for this purpose by the Institutional Review Board (IRB) of the University of Michigan Medical Center indicating that they are aware of the investigational aspects of the treatment and the potential risks.
* Ability to understand and the willingness to sign a written informed consent.
* If a patient is randomized to the RFA arm, but is deemed not to be an anesthesia candidate, he/she will be placed in the non-randomized SBRT cohort.

Inclusion Criteria for non-randomized SBRT arm:

* Patients with renal cell carcinoma less than 8 cm in maximum diameter, patients with metastatic RCC who require local palliation or are progressing through systemic disease, patients who are poor surgical candidates and have tumor location not amenable to RFA, or patients who would prefer a noninvasive means of treatment are eligible for the non-randomized SBRT cohort (Renal cell carcinoma must be pathologically proven).
* There are no limitations based on location of the primary tumor within the kidney.
* Patients must have an ECOG score ≤ 3.
* There is no required minimum renal function (patients will be counseled about the possible need for dialysis, if applicable, just as would be the case for radical or partial nephrectomy).
* Patients must sign an informed consent form approved for this purpose by the Institutional Review Board (IRB) of the University of Michigan Medical Center indicating that they are aware of the investigational aspects of the treatment and the potential risks.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Patients younger than 18 or pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-05; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Spratt, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomized SBRT: Patients who meet eligibility criteria (unilateral primary renal cell carcinoma less than 4 cm in greatest diameter) and are randomized to Stereotactic Body Radiation Therapy (SBRT) will receive SBRT delivered in fractions of 20 Gy, approximately every other day, for a total of three treatments. If the target is deemed too close to organs at risk, 5 fractions of up to 10 Gy per fraction will be prescribed.
  SBRT
- Randomized RFA: Patients who meet eligibility criteria (unilateral primary renal cell carcinoma less than 4 cm in greatest diameter) and are randomized to Radiofrequency Ablation (RFA) will receive RFA.
  RFA
- Non-Randomized SBRT: Patients with renal cell carcinoma's greater than or equal to 4 cm in diameter, and up to 8 cm in diameter, may be placed in the non-randomized stereotactic body radiation therapy arm. Patients with tumors not amenable to RFA, those with metastatic disease, and those who elect a noninvasive means of treatment will also be eligible to receive treatment in the non-randomized SBRT cohort.
  SBRT
Period: Overall Study
Arm/Group | Randomized SBRT | Randomized RFA | Non-Randomized SBRT
Started | 1 | 0 | 3
Completed | 1 | 0 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized SBRT | Randomized RFA | Non-Randomized SBRT | Total
Number analyzed (Participants) | 1 | 0 | 3 | 4
Age, Continuous [Mean (Full Range); unit: years] | 87 [87 to 87] |  | 66 [51 to 87] | 71.25 [51 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 1 | 1
  Male | 1 |  | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Local Control of Disease
Description: On imaging, local control will be defined as when the treated lesion shows no enhancement.
Time Frame: 12 months
Population: Due to changes in the planned scanning procedure during the trial, and feasibility for patients to undergo a diagnostic biopsy and baseline imaging and following imaging requiring contrast was deemed not possible, the trial close secondary to poor accrual and patients were unable to be followed per protocol (data points not captured).
Arm/Group | Randomized SBRT | Randomized RFA | Non-Randomized SBRT
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Cumulative Incidence of Grade 2 and Greater Toxicities
Description: The number of patients reporting grade 2 and greater toxicities (for this trial the Common Terminology Criteria for Adverse Events or CTCAE was used).
Time Frame: up to 30 days after the last study treatment
Population: Although no patients reported toxicity, the trial had poor accrual and patients were unable to be followed per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized SBRT | Randomized RFA | Non-Randomized SBRT
Number analyzed (Participants) | 1 | 0 | 3
Participants | 0 | 0 | 0

3. Secondary Outcome: Difference in Quality of Life (QOL) Scores Between SBRT and RFA Treatment Arms
Description: QOL scores will be summarized descriptively by treatment at each time point using the Convalescence and Recovery Evaluation (CARE) and SF-12 quality of life assessments . Any differences between treatment groups will be tested in the context of a general linear model with terms for treatment, time, treatment time and possibly other patient level covariates that might explain QOL.
Time Frame: Pre-study, last day of treatment; 1, 3, 6, 12, 18, 24 and 36 months post treatment
Population: as for outcome 1
Arm/Group | Randomized SBRT | Randomized RFA | Non-Randomized SBRT
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Difference in Patient Time Away (Measured in Days) Between SBRT and RFA Treatment Arms
Description: Patient time away from work/home secondary to treatment will be captured via patient questionnaire as a number of days and will be summarized descriptively by treatment group. Any differences between treatment groups will be tested by a two-sample t-test or nonparametric Mann-Whitney test.
Time Frame: Pre-study, last day of treatment; 1, 3, 6, 12, 18, 24 and 36 months post treatment
Population: as for outcome 1
Arm/Group | Randomized SBRT | Randomized RFA | Non-Randomized SBRT
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Metastasis Free Survival Time
Time Frame: 36 months post treatment
Population: as for outcome 1
Arm/Group | Randomized SBRT | Randomized RFA | Non-Randomized SBRT
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Overall Survival Time
Time Frame: 36 months post treatment
Population: as for outcome 1
Arm/Group | Randomized SBRT | Randomized RFA | Non-Randomized SBRT
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Difference in Incidence of Treatment Related Pain Between SBRT and RFA Treatment Arms
Description: All patients will be followed to assess the development of treatment related pain, and resultant usage of analgesics (drug classification and dosage) for treatment related pain. Incidence and severity of pain will be recorded for all patients, using the Common Terminology Criteria for Adverse Events (CTCAE), as will any resultant use of analgesics, and these will be compared between the two arms and analyzed in the non-randomized SBRT cohort.
Time Frame: Pre-study, last day of treatment; 1, 3, 6, 12, 18, 24 and 36 months post treatment
Population: as for outcome 1
Arm/Group | Randomized SBRT | Randomized RFA | Non-Randomized SBRT
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Randomized SBRT | Randomized RFA | Non-Randomized SBRT
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes